CLINICAL TRIAL: NCT02984072
Title: A Randomised Double Blind, Placebo Controlled Study of the Efficacy of Topical Menthol for Pain Relief During Topical Photodynamic Therapy
Brief Title: Menthol for PDT Pain Relief
Acronym: MentholPDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015PQ01
Record Dates: First submitted 2016-11-03; First posted 2016-12-06 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol (Active Comparator): 5% menthol in aqueous cream (Dermacool Forte)
  Interventions: Drug: Menthol
- Placebo (Placebo Comparator): Aqueous cream
  Interventions: Drug: Aqueous Cream

INTERVENTIONS:
Drug: Menthol — Topical menthol in aqueous cream
  Other Names: 5% menthol in aqueous cream
  Arms: Menthol
Drug: Aqueous Cream — placebo
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Topical photodynamic therapy (PDT) is widely used to treat superficial non-melanoma skin cancer (NMSC) and dysplasia, notably actinic keratosis and may also be effective in a range of other dermatological conditions. A major limitation of PDT is pain during irradiation. A lack of knowledge of the mechanism of PDT-induced pain has limited the development of effective approaches for prevention or relief of this adverse effect. The investigators have investigated the possible efficacy of menthol for PDT pain ex vivo and will now study this in a clinical trial. This proposal describes the prospective randomised double blind, placebo controlled clinical trial that will be undertaken to investigate the use of topical menthol for PDT-induced pain relief in patients with actinic keratosis of the face and scalp who will be attending general dermatology and PDT outpatient clinics at Ninewells Hospital, Dundee.

DETAILED DESCRIPTION:
This proposal describes the prospective randomised double blind, placebo controlled clinical trial that will be undertaken to investigate the use of topical menthol for PDT-induced pain relief in patients with actinic keratosis of the face and scalp who will be attending general dermatology and PDT outpatient clinics at Ninewells Hospital, Dundee.

This will be undertaken by comparison of 5% menthol in aqueous cream with aqueous cream as placebo and the primary outcome measures will be pain recorded on a visual analogue scale (VAS) during and up to 24 h after PDT. Secondary outcomes are phototoxicity, assessed by a semi-quantitative scoring system immediately after PDT, fluorescence assessed routinely after cream application and before irradiation and outcome based on clinical assessment three months after PDT and patient evaluation. Patients will be involved in the study from the first visit for PDT until the three-month assessment visit after PDT. Data analysis will be undertaken using within-subject paired analyses as patients act as their own control. Information from this study will inform investigators as to whether topical menthol should be routinely incorporated into PDT treatment regimens in order to reduce pain and increase tolerance of treatment. The information will also provide additional information as to the mechanisms of PDT-induced pain and its possible prevention and/or relief.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Adults >18 years. Target population is men or women ≥50 years (only post-menopausal women)
2. Presence of actinic keratoses (AK) on the face and scalp involving both right and left comparable sites.
3. Free of significant physical abnormalities (e.g. tattoos, dermatoses) in the potential treatment area that may cause difficulty with examination or final evaluation.
4. Able to understand and adhere to protocol requirements.

Exclusion Criteria:

1. Unable to give written informed consent.
2. Allergy to menthol, aqueous cream or excipients
3. Participation in a drug trial or other interventional study within 30 days of recruitment to this study
4. Pre-menopausal women, pregnancy, breast feeding, planning to conceive
5. Chronic pain

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Pain immediately after PDT assessed by VAS score | 24h
  pain immediately after and at 3, 6 and 24 h after PDT assessed by VAS score

SECONDARY OUTCOMES:
Clearance: clear/partially clear/not clear - clinical assessment visually and by palpation | 3 months after treatment
  Clearance (CR), partial clearance (PR) or no clearance (NR) will be recorded on each side in each participant
Erythema (redness) (none/mild/moderate/severe) | Immediately after PDT
  Erythema grading (none/mild/moderate/severe) will be recorded on each side in each participant
fluorescence assessed as none/mild/moderate/strong using Wood's light examination | Immediately before and after PDT
  Fluorescence of each side in each participant will be recorded
patient preference - preferred right or left side or no preference | 24h
  patient questionnaire completed at home and returned in SAE
swelling | immediately after PDT
  Swelling present or absent will be recorded on each side in each patient
Exudation | immediately after PDT
  Exudation present or absent will be recorded on each side in each patient
urticaria | immediately after PDT
  Urticaria present or absent will be recorded on each side in each patient

OTHER OUTCOMES:
Blinding - patient will be asked which side they think the menthol was used on or if they do not know | 24h
  patient questionnaire completed at home and returned in SAE

CONTACTS AND LOCATIONS:
Overall Officials: Sally H Ibbotson, MBChB, MD, Principal Investigator — University of Dundee
Locations (1):
- Ninewells Hospital and medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Findings of study will be shared through peer reviewed publications and presentations, although individual participant data not disclosed

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT02984072/Prot_SAP_000.pdf